CLINICAL TRIAL: NCT02721693
Title: COPD, Physical Exercise and Troponin T
Brief Title: Troponin T in Chronic Obstructive Pulmonary Disease (COPD) Patients After Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Responsible Party: Principal Investigator, Anne Helene Edvardsen, Head of Out Patient and Laboratory Department, Researcher, LHL Helse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/23140
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: COPD; Myocardial Diseases
Keywords: Troponin; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiomyopathies; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treadmill exercise test (Experimental): Patients are subjected to an incremental Cardiopulmonary Exercise Test to exhaustion
  Interventions: Device: Treadmill exercise test

INTERVENTIONS:
Device: Treadmill exercise test — Patients are subjected to an incremental exercise test to exhaustion on a treadmill

SUMMARY:
The primary purpose of the study is to investigate if physical exercise is associated with myocardial damage, expressed by elevated troponin T, in patients with COPD.

DETAILED DESCRIPTION:
Patients with COPD will perform a cardiopulmonary exercise test (CPET) on treadmill until exhaustion, 8-12 minutes. Venous blood will be drawn before exercise test and 15 minutes, 3 hours and 24 hours after test for analysis of high sensitive Cardiac troponin T (hs-cTnT). The investigators will also measure arterial bloodgas, oxygen uptake, carbon dioxide consumption, ventilation, blood pressure, ECG, heart rate and ask for dyspnea-score.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* GOLD 2-4
* BODE-index ≥ 2
* Referred by physician to a CPET

Exclusion Criteria:

* Other serious pulmonary diseases (e.g. cancer, sarcoidosis, restrictive pulmonary diseases)
* Chronic heart disease with unstable angina or myocardial infarction ≤ 3 months prior to inclusion
* Percutaneous coronary intervention (PCI)
* Hypertension that is not controlled

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Troponin T concentration 3 h | 3 h

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Edvardsen, PhD, Principal Investigator — LHL Helse
Locations (1):
- LHL-klinikkene, Hakadal, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No